CLINICAL TRIAL: NCT02155972
Title: The Safety and Effectiveness of Probiotic Supplementation on Bipolar Depression: a Proof of Concept Randomized Controlled Trial
Brief Title: The Safety and Effectiveness of Probiotic Supplementation on Bipolar Depression
Acronym: ALIGN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated because of inability to recruit the needed number of participants
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Valerie Taylor, Psychiatrist in Chief, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 179489
Record Dates: First submitted 2014-05-28; First posted 2014-06-04 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Bipolar Depression
Keywords: Bipolar; Depression; Probiotic; ALIGN; HAMD; STAI; YMRS; CGI; SDS; WHOQOL-BREF; C-SSRS; TSES
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive either ALIGN (probiotic) or Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifidobacterium infantis (Active Comparator): Bifidobacterium infantis (Align) 10.00 million cfu capsule once daily
  Interventions: Dietary Supplement: Bifidobacterium infantis
- Placebo (Placebo Comparator): Placebo capsule once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium infantis — Probiotic supplement
  Other Names: ALIGN
  Arms: Bifidobacterium infantis
Other: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
This is an 8-week randomized, double-blind placebo-controlled proof of concept study assessing the combination of a mood stabilizer + Align in the treatment of participants with a bipolar depressive episode. The study has two treatment arms: mood stabilizer plus placebo and mood stabilizer plus Align.

The dose of mood stabilizer will be in accordance with clinical practice guidelines and the dose for Align will be 1 capsule per day as per appropriate product dosing.

DETAILED DESCRIPTION:
Depression has emerged as the major challenge for short- and long-term management of bipolar disorder; new treatments are needed to help control this illness. Studies indicate that probiotics in the stomach improves mood and reduces anxiety symptoms lending further support to the notion that probiotic bacteria positively influence emotional states. We propose to evaluate the effectiveness of the combination of mood stabilizer and Align, a probiotic as compared to mood stabilizer monotherapy.

The primary goal of this feasibility study is to determine the safety and tolerability of Align as an add on to accepted monotherapy treatment in BD. Secondary Objective:1)To evaluate the effectiveness of the combination of mood stabilizer + Align compared to mood stabilizer monotherapy in treatment of BD. 2) to determine if Align +mood stabilizer combination will reduce anxiety symptoms.

An 8-week randomized, double-blind placebo-controlled proof of concept study assessing the combination a mood stabilizer + Align in the treatment of patients with an bipolar depressive episode. The study has two treatment arms: mood stabilizer + placebo and mood stabilizer + Align. Participants will be assessed & administered study scales at screening, baseline & weeks 2,4,6 and 8. the dose for mood stabilizer will be in accordance with clinical practice guidelines and Align - 1 capsule/day.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the nature of the study and have agreed to and are able to read, review, and sign the informed consent form. The informed consent document will be written in English, therefore the volunteer must have the ability to read and communicate in English
* Male and Female participants 18 - 65 years of age ,inclusive, at the time of screening
* Demonstrates a diagnosis of bipolar depression (type I or II) according to the Mini International Neuropsychiatric interview (MINI)
* Is not hospitalized or institutionalized (outpatient) at the time of screening
* Have been on a stable (unchanged) and adequate dose of one of the permissible medications for at least 8 weeks prior to screening (lithium, valproate/divalproex, carbamazepine, lamotrigine, quetiapine/quetiapine XR, olanzapine, or risperidone)
* Demonstrates a maximum HAM-D score of 24 at screening and baseline visits
* Female participants Must:

Not be breast feeding Not be pregnant or seeking to get pregnant during the course of this study. Be menopausal or using an acceptable method of birth control (implants, injectables, combined oral contraceptives, IUDs, sexual abstinence or a vasectomized partner)

Exclusion Criteria:

* Demonstrates or reports a history of any of the DSM-IV criteria for classification of substance abuse/dependence disorders in the past year.
* Demonstrates the presence of active eating disorders, schizophrenia or schizoaffective disorder
* Demonstrates current psychotic symptoms
* Demonstrates a Young Mania Rating Scale (YMRS) score of >12 at screening
* Demonstrates active suicidality based on the C-SSR scale
* Reports using any potent cytochrome P450 inhibitors (such as chloramphenicol, antifungal agents) during the 14 days prior to screening
* Reports a history of electroconvulsive therapy (ECT) during the 90 days prior to screening
* Reports using Align or any other probiotic supplement within the last year prior to screening
* Reports a history of allergic response(s) to components of Align (such as Bifidobacterioum), or any other related drug.
* Reports a presence or history of any medical conditions that would affect drug pharmacokinetics (gastrointestinal conditions such as chroris or colitus).
* Reports a history of any immunocompromising condition (such as HIV, lymphoma, patients undergoing long-term corticosteroid treatment)
* Currently experiencing nausea, fever, vomiting, bloody diarrhea or severe abdominal pain
* Reports use of other natural health products (in addition to probiotics) that affect depression (such as St. Johns Wart, Tryptophan) within the last 6 months prior to screening
* Reports frequent consumption of foods rich in / enriched with probiotics (e.g. yoghurt, drinks, e.t.c).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of Align | 8 weeks
  Tolerability will be assessed using the Toronto Side Effect Scale (TSES). It is a 32-item instrument that is designed to establish incidence, frequency, and severity of central nervous system (CNS), gastrointestinal (GI), and sexual side effects. We will also assess the proportion of participants withdrawing from study due to inadequate control of depressive symptoms or treatment emergent mania

SECONDARY OUTCOMES:
The effectiveness of the combination of mood stabilizer + Align | 8 weeks
  This will be assessed through the change in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score from baseline to the final visit (week 8)
evaluate the combination of mood stabilizer + Align as compared to mood stabilizer monotherapy for participants with bipolar depression with respect to anxiety symptoms and global function/overall improvement | 8 weeks
  Anxiety symptoms will be assessed by looking at the mean change in the State and Trait Anxiety Index (STAI) total score, quality of life will be assessed with the World Health Organization Quality of Life (WHO-QOL) scale and global functioning will be accessed via mean change in the following: Sheehan Disability Scale (SDS) score, the clinical global impressions (CGI) severity of illness score, the CGI-Improvement scale and the CGI Participant Assessment. All measures will be evaluated looking at change from baseline to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Taylor, PhD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's college Research Institute, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bercik P, Verdu EF, Foster JA, Macri J, Potter M, Huang X, Malinowski P, Jackson W, Blennerhassett P, Neufeld KA, Lu J, Khan WI, Corthesy-Theulaz I, Cherbut C, Bergonzelli GE, Collins SM. Chronic gastrointestinal inflammation induces anxiety-like behavior and alters central nervous system biochemistry in mice. Gastroenterology. 2010 Dec;139(6):2102-2112.e1. doi: 10.1053/j.gastro.2010.06.063. Epub 2010 Jun 27. PMID 20600016
- [Background] Cryan JF, O'Mahony SM. The microbiome-gut-brain axis: from bowel to behavior. Neurogastroenterol Motil. 2011 Mar;23(3):187-92. doi: 10.1111/j.1365-2982.2010.01664.x. PMID 21303428
- [Background] Forsythe P, Sudo N, Dinan T, Taylor VH, Bienenstock J. Mood and gut feelings. Brain Behav Immun. 2010 Jan;24(1):9-16. doi: 10.1016/j.bbi.2009.05.058. Epub 2009 May 28. PMID 19481599
- [Background] Rhee SH, Pothoulakis C, Mayer EA. Principles and clinical implications of the brain-gut-enteric microbiota axis. Nat Rev Gastroenterol Hepatol. 2009 May;6(5):306-14. doi: 10.1038/nrgastro.2009.35. PMID 19404271
- [Background] Sudo N, Chida Y, Aiba Y, Sonoda J, Oyama N, Yu XN, Kubo C, Koga Y. Postnatal microbial colonization programs the hypothalamic-pituitary-adrenal system for stress response in mice. J Physiol. 2004 Jul 1;558(Pt 1):263-75. doi: 10.1113/jphysiol.2004.063388. Epub 2004 May 7. PMID 15133062
- [Background] Neufeld KM, Kang N, Bienenstock J, Foster JA. Reduced anxiety-like behavior and central neurochemical change in germ-free mice. Neurogastroenterol Motil. 2011 Mar;23(3):255-64, e119. doi: 10.1111/j.1365-2982.2010.01620.x. Epub 2010 Nov 5. PMID 21054680
- [Background] Diaz Heijtz R, Wang S, Anuar F, Qian Y, Bjorkholm B, Samuelsson A, Hibberd ML, Forssberg H, Pettersson S. Normal gut microbiota modulates brain development and behavior. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3047-52. doi: 10.1073/pnas.1010529108. Epub 2011 Jan 31. PMID 21282636
- [Background] Lyte M, Li W, Opitz N, Gaykema RP, Goehler LE. Induction of anxiety-like behavior in mice during the initial stages of infection with the agent of murine colonic hyperplasia Citrobacter rodentium. Physiol Behav. 2006 Oct 30;89(3):350-7. doi: 10.1016/j.physbeh.2006.06.019. Epub 2006 Aug 2. PMID 16887154
- [Background] Goehler LE, Gaykema RP, Opitz N, Reddaway R, Badr N, Lyte M. Activation in vagal afferents and central autonomic pathways: early responses to intestinal infection with Campylobacter jejuni. Brain Behav Immun. 2005 Jul;19(4):334-44. doi: 10.1016/j.bbi.2004.09.002. PMID 15944073
- [Background] Bravo JA, Forsythe P, Chew MV, Escaravage E, Savignac HM, Dinan TG, Bienenstock J, Cryan JF. Ingestion of Lactobacillus strain regulates emotional behavior and central GABA receptor expression in a mouse via the vagus nerve. Proc Natl Acad Sci U S A. 2011 Sep 20;108(38):16050-5. doi: 10.1073/pnas.1102999108. Epub 2011 Aug 29. PMID 21876150
- [Background] Judd LL, Akiskal HS, Schettler PJ, Endicott J, Maser J, Solomon DA, Leon AC, Rice JA, Keller MB. The long-term natural history of the weekly symptomatic status of bipolar I disorder. Arch Gen Psychiatry. 2002 Jun;59(6):530-7. doi: 10.1001/archpsyc.59.6.530. PMID 12044195
- [Background] Judd LL, Akiskal HS, Schettler PJ, Coryell W, Endicott J, Maser JD, Solomon DA, Leon AC, Keller MB. A prospective investigation of the natural history of the long-term weekly symptomatic status of bipolar II disorder. Arch Gen Psychiatry. 2003 Mar;60(3):261-9. doi: 10.1001/archpsyc.60.3.261. PMID 12622659
- [Background] Gitlin MJ, Mintz J, Sokolski K, Hammen C, Altshuler LL. Subsyndromal depressive symptoms after symptomatic recovery from mania are associated with delayed functional recovery. J Clin Psychiatry. 2011 May;72(5):692-7. doi: 10.4088/JCP.09m05291gre. Epub 2010 Jun 29. PMID 20673560
- [Background] Post RM, Denicoff KD, Leverich GS, Altshuler LL, Frye MA, Suppes TM, Rush AJ, Keck PE Jr, McElroy SL, Luckenbaugh DA, Pollio C, Kupka R, Nolen WA. Morbidity in 258 bipolar outpatients followed for 1 year with daily prospective ratings on the NIMH life chart method. J Clin Psychiatry. 2003 Jun;64(6):680-90; quiz 738-9. doi: 10.4088/jcp.v64n0610. PMID 12823083
- [Background] Post RM, Leverich GS, Nolen WA, Kupka RW, Altshuler LL, Frye MA, Suppes T, McElroy S, Keck P, Grunze H, Walden J; Stanley Foundation Bipolar Network. A re-evaluation of the role of antidepressants in the treatment of bipolar depression: data from the Stanley Foundation Bipolar Network. Bipolar Disord. 2003 Dec;5(6):396-406. doi: 10.1046/j.1399-5618.2003.00065.x. PMID 14636363
- [Background] Joffe RT, MacQueen GM, Marriott M, Trevor Young L. A prospective, longitudinal study of percentage of time spent ill in patients with bipolar I or bipolar II disorders. Bipolar Disord. 2004 Feb;6(1):62-6. doi: 10.1046/j.1399-5618.2003.00091.x. PMID 14996142
- [Background] Gaykema RP, Goehler LE, Lyte M. Brain response to cecal infection with Campylobacter jejuni: analysis with Fos immunohistochemistry. Brain Behav Immun. 2004 May;18(3):238-45. doi: 10.1016/j.bbi.2003.08.002. PMID 15050651
- [Background] Goehler LE, Park SM, Opitz N, Lyte M, Gaykema RP. Campylobacter jejuni infection increases anxiety-like behavior in the holeboard: possible anatomical substrates for viscerosensory modulation of exploratory behavior. Brain Behav Immun. 2008 Mar;22(3):354-66. doi: 10.1016/j.bbi.2007.08.009. Epub 2007 Oct 24. PMID 17920243
- [Background] Li W, Dowd SE, Scurlock B, Acosta-Martinez V, Lyte M. Memory and learning behavior in mice is temporally associated with diet-induced alterations in gut bacteria. Physiol Behav. 2009 Mar 23;96(4-5):557-67. doi: 10.1016/j.physbeh.2008.12.004. Epub 2008 Dec 24. PMID 19135464
- [Background] Culligan EP, Hill C, Sleator RD. Probiotics and gastrointestinal disease: successes, problems and future prospects. Gut Pathog. 2009 Nov 23;1(1):19. doi: 10.1186/1757-4749-1-19. PMID 19930635
- [Background] Verdu EF. Probiotics effects on gastrointestinal function: beyond the gut? Neurogastroenterol Motil. 2009 May;21(5):477-80. doi: 10.1111/j.1365-2982.2009.01297.x. PMID 19432946
- [Background] Camilleri M. Probiotics and irritable bowel syndrome: rationale, putative mechanisms, and evidence of clinical efficacy. J Clin Gastroenterol. 2006 Mar;40(3):264-9. doi: 10.1097/00004836-200603000-00020. PMID 16633134
- [Background] Sullivan A, Nord CE. Probiotics and gastrointestinal diseases. J Intern Med. 2005 Jan;257(1):78-92. doi: 10.1111/j.1365-2796.2004.01410.x. PMID 15606379
- [Background] Gareau MG, Jury J, MacQueen G, Sherman PM, Perdue MH. Probiotic treatment of rat pups normalises corticosterone release and ameliorates colonic dysfunction induced by maternal separation. Gut. 2007 Nov;56(11):1522-8. doi: 10.1136/gut.2006.117176. Epub 2007 Mar 5. PMID 17339238
- [Background] Eutamene H, Bueno L. Role of probiotics in correcting abnormalities of colonic flora induced by stress. Gut. 2007 Nov;56(11):1495-7. doi: 10.1136/gut.2007.124040. PMID 17938427
- [Background] Desbonnet L, Garrett L, Clarke G, Bienenstock J, Dinan TG. The probiotic Bifidobacteria infantis: An assessment of potential antidepressant properties in the rat. J Psychiatr Res. 2008 Dec;43(2):164-74. doi: 10.1016/j.jpsychires.2008.03.009. Epub 2008 May 5. PMID 18456279
- [Background] Girard SA, Bah TM, Kaloustian S, Lada-Moldovan L, Rondeau I, Tompkins TA, Godbout R, Rousseau G. Lactobacillus helveticus and Bifidobacterium longum taken in combination reduce the apoptosis propensity in the limbic system after myocardial infarction in a rat model. Br J Nutr. 2009 Nov;102(10):1420-5. doi: 10.1017/S0007114509990766. Epub 2009 Jun 29. PMID 19563693
- [Background] Rao AV, Bested AC, Beaulne TM, Katzman MA, Iorio C, Berardi JM, Logan AC. A randomized, double-blind, placebo-controlled pilot study of a probiotic in emotional symptoms of chronic fatigue syndrome. Gut Pathog. 2009 Mar 19;1(1):6. doi: 10.1186/1757-4749-1-6. PMID 19338686
- [Background] Logan AC, Katzman M. Major depressive disorder: probiotics may be an adjuvant therapy. Med Hypotheses. 2005;64(3):533-8. doi: 10.1016/j.mehy.2004.08.019. PMID 15617861
- [Background] Silk DB, Davis A, Vulevic J, Tzortzis G, Gibson GR. Clinical trial: the effects of a trans-galactooligosaccharide prebiotic on faecal microbiota and symptoms in irritable bowel syndrome. Aliment Pharmacol Ther. 2009 Mar 1;29(5):508-18. doi: 10.1111/j.1365-2036.2008.03911.x. Epub 2008 Dec 2. PMID 19053980
- [Background] Bailey MT, Coe CL. Maternal separation disrupts the integrity of the intestinal microflora in infant rhesus monkeys. Dev Psychobiol. 1999 Sep;35(2):146-55. PMID 10461128
- [Background] Bailey MT, Lubach GR, Coe CL. Prenatal stress alters bacterial colonization of the gut in infant monkeys. J Pediatr Gastroenterol Nutr. 2004 Apr;38(4):414-21. doi: 10.1097/00005176-200404000-00009. PMID 15085020
- [Background] Tannock GW, Savage DC. Influences of dietary and environmental stress on microbial populations in the murine gastrointestinal tract. Infect Immun. 1974 Mar;9(3):591-8. doi: 10.1128/iai.9.3.591-598.1974. PMID 4593471
- [Background] Suzuki K, Harasawa R, Yoshitake Y, Mitsuoka T. Effects of crowding and heat stress on intestinal flora, body weight gain, and feed efficiency of growing rats and chicks. Nihon Juigaku Zasshi. 1983 Jun;45(3):331-8. doi: 10.1292/jvms1939.45.331. No abstract available. PMID 6632469
- [Background] O'Mahony SM, Marchesi JR, Scully P, Codling C, Ceolho AM, Quigley EM, Cryan JF, Dinan TG. Early life stress alters behavior, immunity, and microbiota in rats: implications for irritable bowel syndrome and psychiatric illnesses. Biol Psychiatry. 2009 Feb 1;65(3):263-7. doi: 10.1016/j.biopsych.2008.06.026. Epub 2008 Aug 23. PMID 18723164
- [Background] Goncharova GI, Liz'ko NN, Liannaia AM, Shilov VM, Spitsa TI. [Bifidobacterium flora status of cosmonauts before and after completing space flights]. Kosm Biol Aviakosm Med. 1981;15(3):14-8. Russian. PMID 7289537
- [Background] Klooker TK, Braak B, Painter RC, de Rooij SR, van Elburg RM, van den Wijngaard RM, Roseboom TJ, Boeckxstaens GE. Exposure to severe wartime conditions in early life is associated with an increased risk of irritable bowel syndrome: a population-based cohort study. Am J Gastroenterol. 2009 Sep;104(9):2250-6. doi: 10.1038/ajg.2009.282. Epub 2009 Jun 9. PMID 19513027
- [Background] Fitzgerald P, Cassidy Eugene M, Clarke G, Scully P, Barry S, Quigley Eamonn MM, Shanahan F, Cryan J, Dinan Timothy G. Tryptophan catabolism in females with irritable bowel syndrome: relationship to interferon-gamma, severity of symptoms and psychiatric co-morbidity. Neurogastroenterol Motil. 2008 Dec;20(12):1291-7. doi: 10.1111/j.1365-2982.2008.01195.x. Epub 2008 Sep 24. PMID 18823288
- [Background] Whitehead WE, Palsson O, Jones KR. Systematic review of the comorbidity of irritable bowel syndrome with other disorders: what are the causes and implications? Gastroenterology. 2002 Apr;122(4):1140-56. doi: 10.1053/gast.2002.32392. PMID 11910364
- [Background] Garakani A, Win T, Virk S, Gupta S, Kaplan D, Masand PS. Comorbidity of irritable bowel syndrome in psychiatric patients: a review. Am J Ther. 2003 Jan-Feb;10(1):61-7. doi: 10.1097/00045391-200301000-00014. PMID 12522523
- [Background] Marks DM, Han C, Krulewicz S, Pae CU, Peindl K, Patkar AA, Masand PS. History of depressive and anxiety disorders and paroxetine response in patients with irritable bowel syndrome: post hoc analysis from a placebo-controlled study. Prim Care Companion J Clin Psychiatry. 2008;10(5):368-75. doi: 10.4088/pcc.v10n0504. PMID 19158975
- [Background] Creed F, Ratcliffe J, Fernandes L, Palmer S, Rigby C, Tomenson B, Guthrie E, Read N, Thompson DG; North of England IBS Research Group. Outcome in severe irritable bowel syndrome with and without accompanying depressive, panic and neurasthenic disorders. Br J Psychiatry. 2005 Jun;186:507-15. doi: 10.1192/bjp.186.6.507. PMID 15928362
- [Background] O'Mahony L, McCarthy J, Kelly P, Hurley G, Luo F, Chen K, O'Sullivan GC, Kiely B, Collins JK, Shanahan F, Quigley EM. Lactobacillus and bifidobacterium in irritable bowel syndrome: symptom responses and relationship to cytokine profiles. Gastroenterology. 2005 Mar;128(3):541-51. doi: 10.1053/j.gastro.2004.11.050. PMID 15765388
- [Background] Hamilton-Miller JMT. Probiotics in the Management of Irritable Bowel Syndrome: A Review of Clinical Trials. Microbial Ecology in Health & Disease 2001;13:212-216
- [Background] Kim HJ, Camilleri M, McKinzie S, Lempke MB, Burton DD, Thomforde GM, Zinsmeister AR. A randomized controlled trial of a probiotic, VSL#3, on gut transit and symptoms in diarrhoea-predominant irritable bowel syndrome. Aliment Pharmacol Ther. 2003 Apr 1;17(7):895-904. doi: 10.1046/j.1365-2036.2003.01543.x. PMID 12656692
- [Background] Kim HJ, Vazquez Roque MI, Camilleri M, Stephens D, Burton DD, Baxter K, Thomforde G, Zinsmeister AR. A randomized controlled trial of a probiotic combination VSL# 3 and placebo in irritable bowel syndrome with bloating. Neurogastroenterol Motil. 2005 Oct;17(5):687-96. doi: 10.1111/j.1365-2982.2005.00695.x. PMID 16185307
- [Background] Kajander K, Hatakka K, Poussa T, Farkkila M, Korpela R. A probiotic mixture alleviates symptoms in irritable bowel syndrome patients: a controlled 6-month intervention. Aliment Pharmacol Ther. 2005 Sep 1;22(5):387-94. doi: 10.1111/j.1365-2036.2005.02579.x. PMID 16128676
- [Background] Niv E, Naftali T, Hallak R, Vaisman N. The efficacy of Lactobacillus reuteri ATCC 55730 in the treatment of patients with irritable bowel syndrome--a double blind, placebo-controlled, randomized study. Clin Nutr. 2005 Dec;24(6):925-31. doi: 10.1016/j.clnu.2005.06.001. Epub 2005 Jul 27. PMID 16051399
- [Background] Bauserman M, Michail S. The use of Lactobacillus GG in irritable bowel syndrome in children: a double-blind randomized control trial. J Pediatr. 2005 Aug;147(2):197-201. doi: 10.1016/j.jpeds.2005.05.015. PMID 16126049
- [Background] McCarthy J, O'Mahony L, O'Callaghan L, Sheil B, Vaughan EE, Fitzsimons N, Fitzgibbon J, O'Sullivan GC, Kiely B, Collins JK, Shanahan F. Double blind, placebo controlled trial of two probiotic strains in interleukin 10 knockout mice and mechanistic link with cytokine balance. Gut. 2003 Jul;52(7):975-80. doi: 10.1136/gut.52.7.975. PMID 12801954
- [Background] Duke K, Murphy S, Smith M. Probiotic performance in IBD is not uniform: a multi-strain comparison in the lymphocyte transfer model of enterocolitis. Gastroenterology. 2004;126:A283-A284.
- [Background] Goldstein BI, Kemp DE, Soczynska JK, McIntyre RS. Inflammation and the phenomenology, pathophysiology, comorbidity, and treatment of bipolar disorder: a systematic review of the literature. J Clin Psychiatry. 2009 Aug;70(8):1078-90. doi: 10.4088/JCP.08r04505. Epub 2009 Jun 2. PMID 19497250
- [Background] Brietzke E, Stertz L, Fernandes BS, Kauer-Sant'anna M, Mascarenhas M, Escosteguy Vargas A, Chies JA, Kapczinski F. Comparison of cytokine levels in depressed, manic and euthymic patients with bipolar disorder. J Affect Disord. 2009 Aug;116(3):214-7. doi: 10.1016/j.jad.2008.12.001. Epub 2009 Feb 28. PMID 19251324
- [Background] Guloksuz S, Cetin EA, Cetin T, Deniz G, Oral ET, Nutt DJ. Cytokine levels in euthymic bipolar patients. J Affect Disord. 2010 Nov;126(3):458-62. doi: 10.1016/j.jad.2010.04.027. PMID 20537397
- [Background] Kauer-Sant'Anna M, Kapczinski F, Andreazza AC, Bond DJ, Lam RW, Young LT, Yatham LN. Brain-derived neurotrophic factor and inflammatory markers in patients with early- vs. late-stage bipolar disorder. Int J Neuropsychopharmacol. 2009 May;12(4):447-58. doi: 10.1017/S1461145708009310. Epub 2008 Sep 4. PMID 18771602
- [Background] Padmos RC, Van Baal GC, Vonk R, Wijkhuijs AJ, Kahn RS, Nolen WA, Drexhage HA. Genetic and environmental influences on pro-inflammatory monocytes in bipolar disorder: a twin study. Arch Gen Psychiatry. 2009 Sep;66(9):957-65. doi: 10.1001/archgenpsychiatry.2009.116. PMID 19736352
- [Background] Desbonnet L, Garrett L, Clarke G, Kiely B, Cryan JF, Dinan TG. Effects of the probiotic Bifidobacterium infantis in the maternal separation model of depression. Neuroscience. 2010 Nov 10;170(4):1179-88. doi: 10.1016/j.neuroscience.2010.08.005. Epub 2010 Aug 6. PMID 20696216
- [Background] Baldessarini RJ, Tondo L. Suicide risk and treatments for patients with bipolar disorder. JAMA. 2003 Sep 17;290(11):1517-9. doi: 10.1001/jama.290.11.1517. No abstract available. PMID 13129995
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Spielberger CD. Manual for the State-Trait Anxiety Inventory. Corsini Encyclopedia of Psychology. 1. Palo Alto, CA: Consulting Psychologists Press; 1983
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Guy W. Global Impression Scale. ECDEU Assessment Manual for Psychopharmacology-Revised. 1976.
- [Background] Arbuckle R, Frye MA, Brecher M, Paulsson B, Rajagopalan K, Palmer S, Degl' Innocenti A. The psychometric validation of the Sheehan Disability Scale (SDS) in patients with bipolar disorder. Psychiatry Res. 2009 Jan 30;165(1-2):163-74. doi: 10.1016/j.psychres.2007.11.018. Epub 2008 Nov 29. PMID 19042030
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Bartram AK, Lynch MD, Stearns JC, Moreno-Hagelsieb G, Neufeld JD. Generation of multimillion-sequence 16S rRNA gene libraries from complex microbial communities by assembling paired-end illumina reads. Appl Environ Microbiol. 2011 Jun;77(11):3846-52. doi: 10.1128/AEM.02772-10. Epub 2011 Apr 1. PMID 21460107
- [Background] American Psychiatric Association. Practice guideline for the treatment of patients with bipolar disorder (revision). Am J Psychiatry. 2002 Apr;159(4 Suppl):1-50. No abstract available. PMID 11958165
- [Background] Goodwin GM; Consensus Group of the British Association for Psychopharmacology. Evidence-based guidelines for treating bipolar disorder: recommendations from the British Association for Psychopharmacology. J Psychopharmacol. 2003 Jun;17(2):149-73; discussion 147. doi: 10.1177/0269881103017002003. PMID 12870562
- [Background] Royal Australian and New Zealand College of Psychiatrists Clinical Practice Guidelines Team for Bipolar Disorder. Australian and New Zealand clinical practice guidelines for the treatment of bipolar disorder. Aust N Z J Psychiatry. 2004 May;38(5):280-305. doi: 10.1080/j.1440-1614.2004.01356.x. PMID 15144505
- [Background] Calabrese JR, Kasper S, Johnson G, Tajima O, Vieta E, Yatham LN, Young AH. International Consensus Group on Bipolar I Depression Treatment Guidelines. J Clin Psychiatry. 2004 Apr;65(4):571-9. No abstract available. PMID 15119923
- [Background] Suppes T, Dennehy EB, Hirschfeld RM, Altshuler LL, Bowden CL, Calabrese JR, Crismon ML, Ketter TA, Sachs GS, Swann AC; Texas Consensus Conference Panel on Medication Treatment of Bipolar Disorder. The Texas implementation of medication algorithms: update to the algorithms for treatment of bipolar I disorder. J Clin Psychiatry. 2005 Jul;66(7):870-86. doi: 10.4088/jcp.v66n0710. PMID 16013903
- [Background] Kunz M, Cereser KM, Goi PD, Fries GR, Teixeira AL, Fernandes BS, Belmonte-de-Abreu PS, Kauer-Sant'Anna M, Kapczinski F, Gama CS. Serum levels of IL-6, IL-10 and TNF-alpha in patients with bipolar disorder and schizophrenia: differences in pro- and anti-inflammatory balance. Braz J Psychiatry. 2011 Sep;33(3):268-74. doi: 10.1590/s1516-44462011000300010. PMID 21971780